CLINICAL TRIAL: NCT03156725
Title: Iron Absorption From Iron-enriched Aspergillus Oryzae is Similar to Ferrous Sulfate
Brief Title: Assessment of Iron Absorption From Aspergillus Oryzae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Dr. Manju B. Reddy, Professor, Iowa State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: HIFS study
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Iron Bioavailability
Keywords: Iron Bioavailability; hepcidin; ferritin; iron absorption; iron status
MeSH Terms: interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Subjects were two meals on two consecutive days with the stable isotopes.
Who Masked: Participant
Masking Description: When 57Fe was added to a meal an empy capsule was consumed by the subjects. 58Fe and natutal abundace iron associated with A. oryzae was consumed in capsule form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous Sulfate (Experimental): The ferrous sulfate group was required to consume a test containing ferrous sulfate (10 mg of 57Fe). Participants received a meal containing 17.6 g egg albumin, 45 g corn syrup solids, 17.5 g corn oil, 6 ml vanilla extract, and 100 ml of distilled water.
  Interventions: Drug: Ferrous Sulfate
- Aspiron (Experimental): The Asprion group was required to follow the same protocol as the 57Fe experimental group, with the exception of taking A. Oryzae containing (8 mg natural abundace Fe and 2 mg 58Fe. Meals composition was similar to ferrous sulafte group.
  Interventions: Dietary Supplement: Aspiron

INTERVENTIONS:
Drug: Ferrous Sulfate
  Arms: Ferrous Sulfate
Dietary Supplement: Aspiron
  Arms: Aspiron

SUMMARY:
The objective of this study was to compare the absorption of a new iron product, iron enriched Aspergillus oryzae to ferrous sulfate in humans using a double stable-isotope technique.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) remains a health crisis worldwide, especially among productive age women and children. Primarily, inorganic iron salts are being used as iron supplementation to treat IDA and are added to food to improve the nutritional value of the daily diet, however side effects and/or low absorption with diets are a result, limiting the impact on IDA. Sixteen female subject, who were 18-35 years, non-pregnancy, non-anemia with marginal lower iron status (ferritin cut-off value <30ug/L) were recruited in this study. Subjects were randomized to orally consume test meal with stable iron isotopes Fe57 (10mg) in sulfate form and Fe58 (2mg) and 8 mg natural abundance iron in Aspiron, in two visits. Blood samples were collected at baseline and two weeks to assess isotope enrichment and iron status indicators, such as hepcidin and ferritin were measured.

ELIGIBILITY:
Inclusion Criteria:

* Marginal iron status (Serum ferritin <30ug/L)
* BMI in the range 18.5-24.9 kg/m2
* Willing to discontinue vitamin and mineral supplements 2 weeks prior and during the study
* Willing to consume stable iron isotope labelled supplement
* Willing to stop getting blood drawn 2 weeks prior to the study and during the study
* Willing to give multiple blood samples at beginning and end of study

Exclusion Criteria:

* Pregnant
* Lactating
* Smoker
* Anemic (hemoglobin < 120 g/L)
* Has gastro-intestinal disease/condition that can affect absorption
* Allergic to any of the meal components

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2014-09-14 (Actual); Study Completion 2016-06-04 (Actual)

PRIMARY OUTCOMES:
iron absorption | 15 days
  Isotope enrichment in the blood samples

SECONDARY OUTCOMES:
iron status | 15 days
  hepcidin and ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Manju B Reddy, PhD, Principal Investigator — Iowa State University

IPD SHARING:
Plan to Share IPD: No
Publication in a journal